CLINICAL TRIAL: NCT06663215
Title: The Effect of School-Based Bullying Prevention Program on Bullying Victimization, Tendencies and Future Expectations of Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Fatma BOZDAG, Associate Professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HRU-BOZDAG-004
Record Dates: First submitted 2024-10-20; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Bullying
Keywords: peer, bullying, future expectation, bullying education
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- intervention group (Experimental)
  Interventions: Other: School Based Bullying Prevention Program

INTERVENTIONS:
Other: School Based Bullying Prevention Program — Three forms were administered to the adolescents: Personal Information Form, Bullying and Cyberbullying Scale for Adolescents (BCE-A) and Adolescent Future Expectations Scale. Adolescents were included in a school-based bullying prevention program the next day. One month later, the forms were administered again.
  Arms: intervention group

SUMMARY:
The aim of this study is to determine the effect of a school-based bullying prevention program on adolescents' bullying victimization, tendencies and future expectations.

DETAILED DESCRIPTION:
Communication is one of the indispensable elements of human history. With the advancement in technology, the use of the internet, social media, and digital tools such as computers and cell phones has taken an important place in human life. Children and young people use the internet for different activities such as doing educational work, exchanging messages via e-mail, playing online games, shopping, using social networks, watching movies and listening to music. It is reported that the age group with the highest rates of computer and internet use is adolescents and young adults (16-24 and 25-34 age groups). Excessive and problematic use of information technologies and the transfer of relationships to virtual environments can bring about some negative situations that may occur in adolescents such as internet addiction and cyberbullying. Cyberbullying, which is the deliberate and regular use of digital technology such as computers, mobile phones and the internet to harass others, includes concepts such as cyberbullying, cyberbullying and cyber victimization. Bullying, which is a proactive behavioral problem, is a situation in which an individual or group repeatedly exhibits humiliating and aggressive behaviors to an individual or group that is relatively weaker than themselves. Bullying and cyberbullying faced by adolescents have become an important problem worldwide.The aim of this study is to determine the effect of a school-based bullying prevention program on adolescents' bullying victimization, tendencies and future expectations.

ELIGIBILITY:
Inclusion Criteria:

* Studying at Şanlıurfa Eyyübiye Atatürk Anatolian High School and agree to participate in the research

Exclusion Criteria:

* not meeting inclusion criteria

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-02 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
bullying tendency | 1 month
  Scores from the Bullying and Cyberbullying Scale for Adolescents
bullying victimization | 1 month
  Scores from the Bullying and Cyberbullying Scale for Adolescents

SECONDARY OUTCOMES:
Future prospects | 1 month
  Scores from the Adolescent Future Expectations Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma Bozdağ, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No